CLINICAL TRIAL: NCT02748928
Title: Clinical Study to Evaluate the Safety and Efficacy of the UltraShape Power Device Using the U-Sculpt Power Transducer for Abdominal Fat and Circumference Reduction
Brief Title: UltraShape Power for Abdominal Fat and Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF21621
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Excess Abdominal Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UltraShape Power treatment to abdomen (Experimental): Eligible subjects will receive 3 treatments, 2 weeks interval, with the UltraShape Power device according to the study protocol and user manual.
  The subject will return for 3 follow up visits: four weeks (4wk FU), eight weeks (8wk FU) and 12 weeks (12wk FU) after the last treatment, for total expected study duration of 16 weeks
  Interventions: Device: UltraShape Power

INTERVENTIONS:
Device: UltraShape Power — Tissue selectivity is achieved by a proprietary knowledge of ultrasound parameters ensuring specific destruction of the fat cells only within the target area. All other types of tissue, such as blood vessels, muscles and peripheral nerves remain intact. There are no thermal effects. Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time
  Other Names: UltraShape

SUMMARY:
Prospective, one arm, baseline-controlled, clinical study for the evaluation of the UltraShape Power treatment using the U-Sculpt Power Transducer for non-invasive abdominal fat and circumference reduction.

DETAILED DESCRIPTION:
Up to 120 healthy adult volunteers, seeking noninvasive abdominal fat and circumference reduction, male and females, 18 to 60 years of age from 6 investigational sites. Eligible subjects will receive 3 bi-weekly treatments (2 weeks interval) with the UltraShape Power device utilizing the U-Sculpt Power Transducer according to the study protocol. Subjects will return for 3 follow-up visits: four weeks (4wk FU), eight weeks (8wk FU) and 12 weeks (12wk FU) after the last treatment (Third Treatment).

Each subject will be enrolled for total expected study duration of 16 weeks. Subject's abdominal fat thickness and circumference will be measured at the measurements points and will be assessed at each visit. Additionally, a subject questionnaire will be completed in each follow-up visit (4wk, 8wk and 12wk FU). Finally, photography will be performed under visible light conditions of the front, right, left and back view. Most of the assessments will occur at each of the visits (all treatments and all follow-up visits) to the clinic.

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible to participate in the study if he/she meets all the following inclusion criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects, 18 and 60 years of age at the time of enrollment
3. Fitzpatrick Skin Type I to VI.
4. Fat thickness of at least 1.5 cm in the treated area (measured by calibrated caliper).
5. Body mass index (BMI): BMI between 22 to 30 (normal to overweight, but not obese).
6. If female, not pregnant or lactating, must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e. oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. In addition, negative urine pregnancy test as tested before each treatment and at the last follow-up visit for women with child-bearing potential (e.g. not menopause).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used, de-identified in evaluations, publications and presentations.

Exclusion Criteria:

A subject is not eligible for participation in this study if he or she meets any of the following exclusion criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker or defibrillator, abdominal aortic aneurism
2. Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction
7. Previous body contouring procedures in the treatment area within 12 months
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
9. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
10. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
11. Very poor skin quality (i.e., severe laxity)
12. Abdominal wall diastasis or hernia on physical examination
13. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
14. Obesity (BMI above 30)
15. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
16. Unstable weight within the last 6 months (i.e., ± 3 percent weight change in the prior six months)
17. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration)
18. Fat thickness lower than 2.5 cm after strapping at the treated area.
19. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trials)
20. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruthie Amir, MD, Study Director — Syneron Medical
Locations (8):
- United States (8):
  - Laser Skin Surgery Center of Northern California, Sacramento, California
  - Prana Medical Aesthetics, Jacksonville Beach, Florida
  - Baumann Cosmetic and Research Institute, Inc, Miami, Florida
  - DuPage Medical Group, Naperville, Illinois
  - A Womans Touch Plastic Surgery, Louisville, Kentucky
  - Syneron Candela Institute for Education Clinic, Wayland, Massachusetts
  - Union Square Laser Dermatology, New York, New York
  - Jewell Plastic Surgery, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No
Overall results shared with study investigators.

REFERENCES:
- [Background] Ascher B. Safety and efficacy of UltraShape Contour I treatments to improve the appearance of body contours: multiple treatments in shorter intervals. Aesthet Surg J. 2010 Mar;30(2):217-24. doi: 10.1177/1090820X09360692. PMID 20442099
- [Background] Moreno-Moraga J, Valero-Altes T, Riquelme AM, Isarria-Marcosy MI, de la Torre JR. Body contouring by non-invasive transdermal focused ultrasound. Lasers Surg Med. 2007 Apr;39(4):315-23. doi: 10.1002/lsm.20478. PMID 17457840
- [Background] Chang SL, Huang YL, Lee MC, Chang CH, Lin YF, Cheng CY, Hu S. Long-term follow-up for noninvasive body contouring treatment in Asians. Lasers Med Sci. 2016 Feb;31(2):283-7. doi: 10.1007/s10103-015-1852-0. Epub 2015 Dec 29. PMID 26714982

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated and Untreated Abdomen: Circumference and fat thickness reduction of abdomen after Ultrashape treatments (three treatments with U-sculpt Power transducer Isppa 660 W/cm^2)
Period: Overall Study
Arm/Group | Treated and Untreated Abdomen
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treated and Untreated Abdomen: Circumference and fat thickness measurements of abdomen before and after Ultrashape treatments of the same subjects
Arm/Group | Treated and Untreated Abdomen
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 62
Fat Thickness [Mean (Standard Deviation); unit: millimeter] | 31.36 (6.44)
Midline Circumference [Mean (Standard Deviation); unit: centimeter] | 92.14 (7.86)

OUTCOME MEASURES:

1. Primary Outcome: Change in Abdominal Fat Thickness Compared to Baseline as Measured by Ultrasound
Description: Abdominal fat thickness change post UltraShape treatments at 12 weeks follow-up (12wk FU) after final treatment versus baseline
Time Frame: Baseline and 16 weeks (4 weeks treatment + 12 week follow up)
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Treated Abdomen: Subjects treated on the abdomen with Ultrashape ultrasound treatments
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 62
percentage change | -10.5 (11)

2. Secondary Outcome: Change in Abdominal Fat Thickness Compared to Baseline as Measured by Ultrasound
Description: Abdominal fat thickness change as measured by ultrasound post UltraShape Power treatments at 4-week, 8-week and 12-week (from baseline visit) versus baseline
Time Frame: Baseline and at 4, 8, and 12 weeks (from baseline visit)
Population: One participant did not attend the 4 week FU (8 weeks from baseline visit) and three participants did not attend the 8 weeks FU (12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 62
percentage change
  Fat thickness change at 4 weeks | -3.2 (8.2)
  Fat thickness change at 8 weeks: number analyzed (Participants) | 61
  Fat thickness change at 8 weeks | -4.3 (8.4)
  Fat thickness change at 12 weeks: number analyzed (Participants) | 59
  Fat thickness change at 12 weeks | -7.0 (9.3)

3. Secondary Outcome: Change in Abdominal Circumference Compared to Baseline
Description: Abdominal circumference change post UltraShape Power treatments
Time Frame: Baseline and at 4, 8, 12 and 16 weeks (from baseline visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 62
centimeter
  Abdominal circumference change at 4 weeks | -1.03 (2.19)
  Abdominal circumference change at 8 weeks: number analyzed (Participants) | 61
  Abdominal circumference change at 8 weeks | -1.29 (2.64)
  Abdominal circumference change at 12 weeks: number analyzed (Participants) | 59
  Abdominal circumference change at 12 weeks | -1.70 (2.52)
  Abdominal circumference change at 16 weeks | -2.26 (2.70)

4. Secondary Outcome: Number of Investigators Reporting Satisfaction With Participants' Treatment Outcome
Description: Satisfaction assessment will be performed independently by the investigator using a 4-point Likert scale questionnaire from 0 = dissatisfied to 3= very satisfied.
  The values in the data table reflect the number of Investigators who were "satisfied" or "very satisfied" (i.e., "reported a 2 or 3") with Participant Treatment Outcome, as assessed by the questionnaire.
Time Frame: 8, 12 and 16 weeks (from baseline visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Treated Abdomen: Abdomen treated with UltraShape ultrasound treatments
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 62
Participants
  Investigator satisfaction rate at 8 week: number analyzed (Participants) | 61
  Investigator satisfaction rate at 8 week | 44
  Investigator satisfaction rate at 12 week: number analyzed (Participants) | 59
  Investigator satisfaction rate at 12 week | 43
  Investigator satisfaction rate at 16 week | 54

5. Secondary Outcome: Number of Participants Reporting Satisfaction With Treatment Outcome
Description: Satisfaction assessment will be performed independently by the subjects using a 4-point Likert scale questionnaire from 0 = dissatisfied to 3= very satisfied.
  The values in the data table reflect the number of participants who were "satisfied" or "very satisfied" (i.e., "reported a 2 or 3") with Treatment Outcome, as assessed by the questionnaire.
Time Frame: 8, 12 and 16 weeks (from baseline visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 62
Participants
  Subject satisfaction rate at 8 week: number analyzed (Participants) | 61
  Subject satisfaction rate at 8 week | 47
  Subject satisfaction rate at 12 week: number analyzed (Participants) | 59
  Subject satisfaction rate at 12 week | 42
  Subject satisfaction rate at 16 week | 46

6. Secondary Outcome: Pain Scale for Rating Discomfort Associated With Treatment
Description: Comfort assessment will be performed independently by the subjects using a numerical scale (0-no discomfort to 10-Worst possible discomfort). The subjects will answer this questionnaire after each of the three treatments.
Time Frame: Day 0 (1st treatment), at 2 weeks (2nd treatment) and at 4 weeks (3rd treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated Abdomen
Number analyzed (Participants) | 62
score on a scale
  Subject discomfort at first treatment | 0.32 (0.91)
  Subject discomfort at second treatment | 0.25 (0.70)
  Subject discomfort at third treatment | 0.17 (0.70)

ADVERSE EVENTS:
Time Frame: Subjects were assessed and followed up for adverse events at each treatment (3 treatments at 2 weeks interval) and at 4 weeks, 8 weeks and 12 weeks after the Ultrashape Power treatment
Arm/Group | Treated Abdomen
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 11/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Abdomen (N=62)
Welts (Skin and subcutaneous tissue disorders) | 9 (9) — Small mild welts
Pruitis / itching (Skin and subcutaneous tissue disorders) | 1 (1) — Itching following treatment
Blanching (Skin and subcutaneous tissue disorders) | 1 (1) — Mild blanching

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT02748928/Prot_SAP_000.pdf